CLINICAL TRIAL: NCT05283291
Title: The Effect of Directed Imagery Technique Applied to Patients Who Have Had Lumbar Disc Herniation Surgery on Patients' Pain, Anxiety, and Sleep Levels: A Randomized Controlled Study
Brief Title: Directed Imagery Technique Applied to Patients Undergoing Lumbar Disc Herniation Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Eda Albayrak, Research Assistant, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ErciyesU-Albayrak-001
Record Dates: First submitted 2022-02-09; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-02

CONDITIONS: Intervertebral Disc Disorder Lumbar With Radiculopathy; Surgical or Other Invasive Procedure on Wrong Patient; Nurse-Patient Relations
Keywords: Directed Imagery Technique; Herniated Disc; ache; anxiety; Sleep
MeSH Terms: conditions — Intervertebral Disc Displacement; Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İmaginary group (Experimental): Expert opinion for the scenario will be taken from a psychologist and a psychiatric nurse.
  The flow of the script; It will start with breathing exercises and continue with the safe place application, after affirming the functionality that is said while in a safe place in the mind, it will be in the form of waking up by turning to the body and returning to the present.
  Headphones will be provided for each patient by the researcher. In the first meeting, the voice recordings will be transferred to the phones of the individuals via the phone in the Neurosurgery Service. Communication with the patient will be provided in accordance with the pandemic rules.
  The audio recording will be played twice, in the evening before the operation and on the evening of the operation day.
  Interventions: Behavioral: Directed Imagery Technique
- Control group (No Intervention): In the routine care applied to the patients, the vitals of the patients are followed, drug treatments are administered and the motor functions of the patients are monitored. In addition, analgesics are routinely administered in the ward for pain and no attempt is made for sleep.

INTERVENTIONS:
Behavioral: Directed Imagery Technique — The sound recording will include a soothing light background music for approximately 30 minutes.
  Imagination will be practiced, starting with the patient's focusing his/her attention on his/her breath, relaxation, and relaxation with the suggestions given in the recording with the accompaniment of relaxing music.
  Arms: İmaginary group

SUMMARY:
The Directed Imagery technique (YIT) is a set of stories that people create by first giving relaxation exercises and then visualizing the symbols given by the practitioner. Guided imagery is based on the understanding that the body and mind are interconnected and that the mind can affect the body. In directed imagery, the person's thoughts and imagination are focused and directed to a specific goal by the practitioner, usually through a sound recording. The directed imagery technique can be effective in solving problems such as pain, stress, fatigue, and anxiety in nursing care.

DETAILED DESCRIPTION:
1. Patients in the control group; Nursing care will be applied according to the routine care protocol of the clinic where the research was conducted.
2. Patients in the experimental group; In addition to the nursing care given according to the routine care protocol of the clinic where the research was conducted, the "imagery method" will be applied four times in total, once before the operation, once on the 1st day, 2nd day and 3rd day after the operation. It will be ensured that the patients to be imaged are in the supine or semifawler position in a comfortable way and listen to the audio recording with headphones.

Before the application, the patient will be told to listen to the audio recording with headphones at the most convenient time of the day for him, in an environment where he will not be disturbed by others, by putting his phone in airplane mode, after giving advance notice to avoid disturbing family members. Headphones will be provided for each patient by the researcher. In the first meeting, the voice recordings will be transferred to the phones of the individuals via the phone in the Neurosurgery Service. Communication with the patient will be provided in accordance with the pandemic rules. In the preoperative period, "Descriptive Information Form", "Operation-Specific Anxiety Scale", "Richard-Campbell Sleep Scale", "Visual Analog Scale (VAS)", "State Anxiety Scale" will be applied to the experimental and control groups before imagery is performed. After the interventions applied to the experimental group are completed, the scales will be re-administered to the individuals in the experimental and control groups.

ELIGIBILITY:
Inclusion Criteria:

1. Those who will undergo lumbar disc hernia surgery
2. Compliant with ASA 1 and 2 classification
3. Preoperative hospitalizations
4. Patients without cognitive clouding
5. Patients who can speak Turkish
6. Patients without hearing and vision problems will be included in the study.

Exclusion Criteria:

1. Those over the age of eighty or under the age of 18
2. Having a psychiatric disease and using medication
3. Having trouble sleeping and taking medication
4. Those who are classified as ASA 3 and above,
5. Those who have laparoscopic surgery,
6. Those with chronic pain, alcohol, drug and substance addiction,
7. Oncological cases,
8. Those with hearing, vision, speech and cognitive dysfunction,
9. Those who do not speak Turkish,
10. People with high anxiety who use anxiolytics
11. Patients who do not accept the procedure will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Preoperative Anxiety Scale | Change: [Time Frame: 3 days: Preoperative assessment (Time 1), morning of surgery day (Time 2)]
  The range of scores that can be taken from the scale is 10-50 points, and high scores reflect high anxiety.
Richards Campbell Sleep Scale | Change: [Time Frame: 3 days: Preoperative assessment (Time 1), morning of the day of surgery (Duration 2), postoperative (Duration 3)
  Each item is evaluated on a chart between 0 and 100 using the visual analog scale technique. A score of "0-25" from the scale indicates "very bad sleep" and a score of "76-100" indicates "very good sleep".
Visual Analog Scale (VAS) | Change: [Time Frame: 3 days: Preoperative assessment (Time 1), morning of the day of surgery (Duration 2), postoperative (Duration 3)
  "0" describes no pain, "100" describes the most unbearable pain. A score of "0-30" indicates mild pain, a score of "31-60" indicates moderate pain, and a score of "61 and above" indicates severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Eda Albayrak, Principal Investigator — TC Erciyes University
Locations (1):
- Eda Albayrak, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.